CLINICAL TRIAL: NCT01501084
Title: Effects of the GLP-1 Exenatide on Intrinsic Brain Activity in Lean and Obese Women
Brief Title: Effects of the GLP-1 Exenatide on Satiety in Lean and Obese Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Amylin Pharmaceuticals, LLC. (Industry)
Responsible Party: Principal Investigator, Lisa Kilpatrick, PhD, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 11-002316
Record Dates: First submitted 2011-12-20; First posted 2011-12-29 (Estimated); Last update posted 2017-11-07 (Actual); Status verified 2017-11

CONDITIONS: Obesity
Keywords: functional MRI; Structural MRI; obesity; resting state networks
MeSH Terms: conditions — Obesity | interventions — Exenatide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exenatide (Active Comparator): Exenatide injection 10 mcg subcutaneous
  Interventions: Drug: Exenatide
- Saline (Placebo Comparator): .2cc SC injection of sterile normal saline
  Interventions: Drug: Normal saline .2cc subcutaneous injection

INTERVENTIONS:
Drug: Exenatide — 10mcg sc (subcutaneous) injection once at one of the 2 MRI visits
  Other Names: Byetta
  Arms: Exenatide
Drug: Normal saline .2cc subcutaneous injection — sterile saline injection
  Arms: Saline

SUMMARY:
Obesity is a major health problem in the US and many Western countries, with more than half of the population being overweight or obese. Yet, despite intense research efforts into the mechanisms underlying obesity and into the development of novel pharmacologic interventions, bariatric surgery, including gastric bypass surgery is the only successful treatment for severe obesity. Mimicking one of the effects of bariatric surgery, e.g. the increased secretion of glucagon-like peptide 1 (GLP-1) could be an effective strategy against obesity.

Obese individuals may be more sensitive to the rewarding aspects of food and less responsive to signals from the gut about actual energy needs. Using functional MRI scanning the investigators plan to examine the effect of Exenatide (a GLP-1 analog known to reduce caloric intake and produce weight loss in both obese and lean individuals) on activity within brain regions/networks involved in reward/motivation and in regulation of energy requirements. The investigators expect the peptide to change the balance between desire to eat for pleasure and the need to eat to maintain homeostasis.

DETAILED DESCRIPTION:
PRIMARY STUDY OBJECTIVE The proposed study aims to address two important questions regarding the mechanisms underlying the weight loss associated with exenatide. The investigators primary study objective is to determine whether Exenatide changes the resting state activity of the brain, and alters the connectivity between brain regions involved in homeostatic and hedonic brain circuits.

SECONDARY STUDY OBJECTIVE The secondary study objective is to determine if/how these changes differ between lean and obese subjects

SIGNIFICANCE Obesity is a major health problem in the US and many Western countries, with more than half of the population being overweight or obese. Yet, despite intense research efforts into the mechanisms underlying obesity and into the development of novel pharmacologic interventions, bariatric surgery, including gastric bypass surgery is the only successful treatment for severe obesity (le Roux, 2006; le Roux, 2007). Mimicking one of the effects of bariatric surgery, e.g. the increased secretion of glucagon-like peptide 1 (GLP-1) could be an effective strategy against obesity (Torekov, 2011).

The impact of gut peptides on the brain in the regulation of ingestive behavior is an area of great interest, since the involved signaling mechanisms may be potential targets for the treatment of obesity. Both endocrine, paracrine and neurocrine (vagal) signaling pathways are involved in gut to brain signaling of nutrient related information (Holst, 2007). Human studies have demonstrated that long acting hormones like leptin and insulin act on brain regions such as the hypothalamus and brainstem, influencing both food intake and response (Ahima, 2010). More short -term gut signals relayed by hormones such as CCK and PYY have also been shown in humans to have an effect on subcortical regions (including the hypothalamus, nucleus tractus solitarius (NTS), pons, thalamus) as well as on cortical regions (middle temporal gyrus, insula and anterior cingulate cortex (ACC) (Ahima, 2010). Whereas CCK infusion in healthy human subjects was found to result in increased activity primarily in homeostatic brain regions (hypothalamus, brainstem), PYY infusions were associated with increased activity in regions of reward-circuits (orbitalfrontal cortex, insula, anterior cingulate cortex). To our knowledge, the central effects of GLP-1 in humans have not been studied. (Ahima, 2010)

HYPOTHESIS

1. Exenatide changes intrinsic activity in the NTS and hypothalamus, and connectivity between NTS and homeostatic and hedonic brain circuits
2. These changes are seen both in lean and in obese subjects
3. Changes in the engagement of brain circuits induced by Exenatide are correlated with increased ratings of satiety following a test meal

METHODS

The study design is a double-blind, placebo controlled, crossover study.

Twenty healthy female subjects between the ages of 18-40 years are needed The subjects will be divided into two age-matched groups of obese and lean women. The ten obese females will have a BMI between 30-35kg/ m2 and the 10 lean females will have a BMI between 19-25kg/m2. All subjects will be asked to participate in the entire protocol of 3 visits. There will be a screening visit to determine eligibility followed by two functional MRI visits where the subject is given a subcutaneous injection (sc) of 10ug of Exenatide (a GLP-1 analog) at one visit and a an injection of saline at the other MRI visit. The choice of female participants is based on the greater prevalence of obesity in women and the longstanding interest of the center's interest in women's health. In order to control for menstrual cycle hormonal fluctuation all participants will be scanned during the follicular phase of the menstrual cycle, for this study defined as the 4th-12th day after starting menstruation.

Screening (Visit 1):

All potential subjects will be asked to complete an initial screening visit approximately 1.5 hours of time. This visit will take place at the Gail and Gerald Oppenheimer Family Center for Neurobiology of Stress at 10833 Le Conte Ave., Los Angeles, CA 90095 Room 47-126. At the beginning of this visit, the subject will be given ample time to read and sign the informed consent. The protocol will be discussed and reviewed with a study MD or RN.

The screening will include a medical history and physical examination. A urine test for pregnancy will also be done. If the pregnancy test is positive the subject will be immediately dropped from participation. Female subjects of child bearing potential will be asked to practice a medically approved birth control method during the study, including the oral contraceptive pill, abstinence, double barrier method (spermicide and condoms), or IUD. A menstrual cycle history will be obtained as part of the medical history and the first day of their last menses will be documented. fMRI visits will be planned during the follicular stage- specifically day 4-12 of their cycle. A 5 cc (1 tsp) blood draw for glucose will be collected. If the non- fasting blood glucose result is more than 200mg/dl the subject will be considered a screen fail. This value was chosen in order to exclude subjects with undiagnosed underlying diabetes.

Subjects will be asked to fill out several behavioral questionnaires: the UCLA bowel symptom questionnaire (BSQ 5.0), the Hospital Anxiety and Depression scale (HAD), the Spielberger State and Trait Anxiety Inventory (STAI-Y1 and Y2) and the MRI safety screening questionnaire; requiring about 20 minutes to complete.

The RN, NP or MD will review the inclusion and exclusion criteria with the subject to determine eligibility.

A brief structured psychological interview (MINI+) will be done to identify any major Axis I psychiatric disorders in DSM-IV and ICD-10, such as anxiety, depression, substance abuse or phobias.

If the subject is eligible and wishes to participate, they will be provided with instructions for the following study visit. As noted this visit will be scheduled during the follicular phase of the individual's menstrual cycle.

Visit 2 MRI scanning visit 1:

This visit will take approximately 2 hours of time. Subject will be asked to fast (except water) for eight hours prior to admission. Eligibility criteria for continuance in the study, including adverse events and any change in medication usage will be reviewed and recorded. The 1st day of last menstrual period will be noted and a urine pregnancy test will be performed. If positive the subject will be removed from study enrollment.

Subjects will be escorted to the CTSI (General clinical research area) and an IV will be placed for the four blood draws. A baseline fasting blood glucose will be done. It needs to be between 65mg/dl and 126mg/dl or the visit will be cancelled. The subject will then be escorted to the UCLA Ahmanson-Lovelace Brain Mapping Center, 660 Charles Young Dr. South, Los Angeles, CA 90095-7085 and prepared for scanning. Subjects will be asked to complete a PROMIS questionnaire prior to scanning to evaluate the previous nights sleep quality (for RSN analysis) and a Fullness Questionnaire (FQ); a visual analog scale used to measure hunger and satiety.

After wanding for metal safety they will be escorted into the MRI chamber. They will be given a synopsis of the study tests and prepared for placement in the scanner. They will be monitored for pulse oximetry and respiratory rate as a measure of autonomic nervous system and as a safety measure (after Exenatide injection) while scanning. These measures will be collected during all functional resting state network (RSN) scans.

Following placement structural scans will be done After the structural scans the subject will undergo a 10-minute resting state (RSN) scan during which then they will be asked to lie still with their eyes closed but not fall asleep.

After that RSN scan, subjects will be partially moved out of the scanner to receive either a subcutaneous injection of 10ug of Exenatide or a 0.5cc injection of saline (placebo) in the upper arm, thigh or abdomen. Randomization will be done by the UCLA research pharmacy where the drug is stored and dispensed. Subject and investigator will blinded to the randomization.

Immediately following the injection the subject will be moved back into the scanner and have a 8.5 minute structural scanner (MP Rage: a three-dimensional, T1-weighted, gradient-echo sequence used for study analysis). Immediately following the MP Rage, the subject will have the second 10-minute RSN scan (10-minutes post drug) with the same RSN instructions. After the second RSN scan is completed the subjects will complete the second Fullness Questionnaire (FQ). This will be presented on the screen via goggles and the answers will be given to the scanner operator via intercom. The subject will then be partially moved out of the scanner for a 1 teaspoon (5cc) blood draw. This serum sample will be for glucose, insulin and exenatide pharmacokinetic.

The subject will then be moved back into the scanner for the third and final 10-minute RSN with the same previous instructions. Immediately following this scan the subject will complete the third FQ and have 1 teaspoon (5cc) of blood drawn for glucose, insulin and Exenatide pharmacokinetic levels.

After scanning, subjects will be taken to the CTSI and provided a full balanced standard meal of 1200 calories. All subjects will have 2 lunch meal choices to choose from (chicken or ham) and will be instructed to "eat until you are full". After the meal, the subject will complete the fourth FQ and a final 5cc blood draw for glucose, insulin and Exenatide PK level. Approximate blood sampling for the whole day will be 1-2 ounces.

All scanning will be done in the morning, between ~9am-12pm, to account for hormonal fluctuation and for fasting comfort of the subject.

Visit 3 MRI scanning Visit 2:

Visit 3 is identical to Visit 2 except the subject will receive the opposite injection. If the subject was randomized to receive 10ug of Exenatide during Visit 2 then she will receive .5cc of saline (placebo) during Visit 3. Otherwise study procedures will be identical.

ELIGIBILITY:
Inclusion Criteria:

1. FEMALES 18 to 40 years of age, inclusive
2. Lean control subjects with BMI's between 19 and 25kg/m2.
3. Obese subjects with BMI's between 30 and 35kg/m2.
4. Willingness to participate in this study as evidenced by a signed, written informed consent form (ICF).
5. Willingness to avoid pregnancy and practice adequate birth control (abstinence, oral contraception, intrauterine devices, implantable devices, or barrier method with spermicide) during the time of study enrollment.
6. Negative urine pregnancy tests at all visits.
7. All subjects must be premenopausal.
8. In the follicular stage of the menstrual cycle, as determined by menstrual history at Visit 2 &3.
9. Ambulatory outpatient (not depending exclusively on a wheelchair for mobility)
10. English is primary oral and written language.
11. Random (non fasting) Blood sugar level < 200mg/dl at screening.
12. Right-handed

Exclusion Criteria

1. Evidence of structural abnormality of the gastrointestinal tract or GI diseases/conditions. Exclusionary GI conditions include but are not limited to: gastrointestinal surgery (exceptions: appendectomy, benign polypectomy, cholecystectomy), pancreatitis, irritable bowel syndrome (IBS), inflammatory bowel disease (IBD), esophagitis (exception: symptom controlled reflux disease), celiac disease, gastrointestinal malignancy or obstruction, functional dyspepsia, peptic ulcer disease, lactose intolerance or any malabsorptive condition.
2. Clinical evidence of cardiovascular, respiratory, renal, hepatic, malignancy, hematologic, neurologic (including regular migraines defined as more than 1 migraine per month), psychiatric or any disease that the PI determines may interfere with safe participation in the study.

   * Very specifically subjects with any history or symptoms of poor glucose control, osteoporosis, diabetes, thyroid, adrenal or other endocrine disorder.
3. Subjects with current psychiatric disorder, or history of such disorder in the past 5 years. This list includes but is not limited to bipolar disorder, alcohol or substance abuse/dependence, suicide attempt or behavior, or presence of anxiety or depression at the time of screening. Poorly controlled anxiety or depression will be determined as a result of MINI + interview by the clinician at screening.
4. Current history of chronic pain.
5. Use of investigational drugs, products or devices within 28 days prior to screen and through study participation.
6. Subjects with current use of any medications/drugs during the study that affect the central nervous system, gastrointestinal motility, autonomic activity or pain sensation, including but not limited to: opiates or other narcotic analgesics, THC, alpha adrenergic receptor antagonists, beta blockers, Ca+ blockers, prokinetics and sympatholytic agents, or antidepressants.
7. Subjects who have used diet aids within the last month.
8. Pregnancy, postpartum within 4 months or breast-feeding
9. Subjects who smoke more than 5 cigarettes per month.
10. Subjects with BMI of less than 20, between 26 and 29 and over 35.
11. Subjects with metal implants, dental retainers, large tattoos (e.g. full arm or back) or claustrophobia; making MRI safety not possible.
12. Any clinically significant abnormalities from the screening medical history or physical examination.
13. Subjects who exercise excessively (more than 8 hours a week on average).
14. Postmenopausal women and/or women who have had oophorectomies.
15. Any other condition that the investigator believes would jeopardize the safety or rights of the subject or would render the subject unable to comply with the study protocol.
16. Subject taking any medications that might interfere or react badly with the GLP-1 agonist: Exenatide
17. Subjects with a non-fasting blood glucose level at > 200 dl/ml.
18. MRI visits with fasting blood sugar < 65 or 126 mg/dl
19. Left handedness

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2011-12; Primary Completion 2012-12 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Resting State networks in the brain | one year
  The proposed study aims to address two important questions regarding the mechanisms underlying the weight loss associated with exenatide. Our primary study objective is to determine whether Exenatide changes the resting state activity of the brain, and alters the connectivity between brain regions involved in homeostatic and hedonic brain circults.

SECONDARY OUTCOMES:
Age and body size differences | one year
  The secondary study objective is to determine if/how these changes differ between lean and obese subjects

CONTACTS AND LOCATIONS:
Overall Officials: Emeran A Mayer, MD/co-PI, Study Director — Oppenheimer Family Center for Neurobiology of Stress at UCLA; Lisa Kilpatrick, PhD, Principal Investigator — Oppenheimer Family Center for Neurobiology of Stress at UCLA
Locations (1):
- UCLA Gail and Gerald Oppenheimer Family Center for Neurobiology of Stress, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes